CLINICAL TRIAL: NCT04485858
Title: Prospective, Open Label, Single Arm, First in Human (FIH) Clinical Study to Assess Safety and Efficacy of the CorNeat Keratoprosthesis for the Treatment of Corneal Blindness
Brief Title: First in Human (FIH) Study to Assess Safety and Efficacy of the CorNeat KPro for the Treatment of Corneal Blindness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: CorNeat Vision Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMS-15012
Record Dates: First submitted 2020-07-08; First posted 2020-07-24 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Corneal Disease; Corneal Opacity; Corneal Injuries
MeSH Terms: conditions — Corneal Diseases; Corneal Opacity; Corneal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CorNeat KPro (Experimental): Intraocular implantation of the CorNeat KPro
  Interventions: Device: CorNeat KPro

INTERVENTIONS:
Device: CorNeat KPro — CorNeat KPro will be implanted into the subject's eye where the optic component snaps into the patient's trephined cornea and is sutured to the eye wall using 3 non-degradable sutures and the skirt component is placed under the conjunctiva

SUMMARY:
Prospective, open label, single arm, First in Human (FIH) clinical study to assess safety and efficacy of the CorNeat Keratoprosthesis, a synthetic cornea, for the treatment of corneal blindness

DETAILED DESCRIPTION:
The objective of this clinical study is to prove the safety and effectiveness of the CorNeat Keratoprosthesis (KPro), a synthetic, artificial cornea for or the treatment of corneal blindness in subjects who are not candidates for traditional corneal transplant.

Ten subjects who are willing to take part in the study will undergo screening examinations to verify their eligibility.

The CorNeat KPro will be implanted unilaterally in eligible subjects. Follow up procedures will be performed at 1 day, 1 week, 1, 2, 3, 6, 9 & 12 months post implantation and will include clinical assessment of the implanted eye using slit-lamp biomicroscopy, intra ocular pressure measurement and ocular imaging. Additionally, subjects' visual acuity will be assessed and recorded throughout the 12 months follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 and ≤ 80 years on the day of screening
* Candidates must have the ability and willingness to attend all scheduled visits and comply with all study procedures
* Keratoprosthesis surgery is indicated in cases when keratoplasty is not a reasonable option or following a verifiable history of prior failed corneal transplantation
* Indications that fall under poor candidate for keratoplasty include but are not limited to: herpetic keratitis, vascularized corneal scar, Ocular Cicatricial Pemphigoid, alkali burn, Steven Johnson Syndrome, and limbal stem cell deficiency
* Pseudophakia
* Adequate tear film and lid function
* Perception of light in all quadrants
* Female patients of childbearing age must have negative pregnancy test at screening and agree to use an effective method of contraception throughout the study

Exclusion Criteria:

* Reasonable chance of success with traditional keratoplasty
* Current retinal detachment
* Connective tissue diseases
* End-stage glaucoma
* History or evidence of severe inflammatory eye diseases (i.e. uveitis, retinitis, scleritis) in one or both eyes within 6 months prior to planned implantation
* History of ocular or periocular malignancy
* History of extensive keloid formation
* Any known intolerance or hypersensitivity to topical anaesthetics, mydriatics, or component of the device
* Signs of current infection, including fever and current treatment with antibiotics
* Severe generalized disease that results in a life expectancy shorter than a year
* Any clinical evidence that the investigator feels would place the subject at increased risk with the placement of the device
* Corneal thickness less than 400 or higher than 1,200 microns in any region of the pachymetry map of the eye intended to be operated
* Currently pregnant or breastfeeding
* Participation in any study involving an investigational drug or device within the past 30 days or 5 half-lives of the drug (whichever longer) or ongoing participation in a study with an investigational drug or device
* Intraoperative complication that would preclude implantation of the study device
* Vulnerable populations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Cincinnati Eye Institute, Edgewood, Kentucky, United States
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - UHN - University Health Network, Toronto, Ontario
- France (2):
  - CHU de Montpellier, Montpellier
  - Hopital Fondation Adolphe de Rothschild, Paris
- Rabin Medical Center - Beilinson, Petah Tikva, Israel
- Netherlands (2):
  - Amsterdam UMC - Location AMC, Amsterdam
  - Maastricht UMC+, Maastricht

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CorNeat KPro
Started | 10
Implantations in Israel, France, Canada | 10
Improved Visual Acuity at Some Point Throughout the Study | 8
VA Improvement at Their Last Follow up Visit They Attended (After 6-24 Months From Surgery) | 4
Completed | 5
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | CorNeat KPro
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: Years] — Aged between 38 and 78 years old.
  Years | 64.6 [38 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  Canada | 5
  Israel | 3
  France | 2
Slit lamp examinations [Number; unit: participants]
  Normal Lids/Lashes/Lacrimal | 5
  Trichiasis Lids/Lashes/Lacrimal | 2
  Tarsorrhaphy Lids/Lashes/Lacrimal | 2
  Ptosis Lids/Lashes/Lacrimal | 1
  Normal conjunctiva | 10
  Mild cornea edema | 1
  Moderate cornea edema | 5
  Severe cornea edema | 4
  AC deep | 8
  AC medium | 1
  No flare | 5
  No Fibrin present | 7
  No cells present | 5
  Normal iris | 5
  Anirdia iris | 1
  Morcher, iris prosthetic | 1
  Normal pupil | 7
  Normal vitreous body | 4
  Pale optic nerve | 1
  Normal macula | 1
  Normal retinal vessels | 2
  Normal retinal periphery | 2
Ocular imaging [Count of Participants; unit: Participants]
  Pachymetry | 7
  AC depth | 3
  AC Morphology | 6
  Location and position of IOL | 5
  Angle Morphology | 7
Pain assessment [Number; unit: participants]
  No or minimal pain (grades 0-2) | 8
  Mild pain (grades 3-4) | 1
  Moderate pain (grades 5-7) | 1
  Severe pain (grades 8-10) | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint as Determined by the Frequency and Severity of All Unanticipated Adverse Device-related Events (UADE)
Description: The frequency and severity of all unanticipated adverse device-related events (UADE) or treatment-related adverse events, during and after implantation of the CorNeat KPro and up to 12 months should be less than SOC
Time Frame: Throughout the 12 months follow up period
Measure: Number; unit: Participants
Arm/Group | CorNeat KPro
Number analyzed (Participants) | 10
Participants | 7

2. Secondary Outcome: Secondary Effectiveness Endpoint - Improvement in BCDVA
Description: Improvement in BCDVA (using ETDRS visual acuity chart, where applicable) compared to baseline
Time Frame: Throughout the 12-months post operation
Measure: Count of Participants; unit: Participants
Arm/Group | CorNeat KPro
Number analyzed (Participants) | 10
Participants | 8

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | CorNeat KPro
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CorNeat KPro (N=10)
Covid 19 Infection (Infections and infestations) | 1
Exposure of implant (Eye disorders) | 1
Flat AC with bleeding (Eye disorders) | 1
Fungal infection in the skirt of artificial cornea (Eye disorders) | 1
Headache (General disorders) | 1
Shallow retinal detachment (Eye disorders) | 1
Dehiscence of prosthesis superiorly (Eye disorders) | 1
Conjunctival retraction with dehiscence of prosthesis & possible corneal epithelial ingrowth (Eye disorders) | 1
Choroidal detachment and exudative detachment (Eye disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CorNeat KPro (N=10)
Metabolic acidosis (Eye disorders) | 1
Retro prosthetic membrane (Eye disorders) | 1 (3)
Exposed synthetic skirt of the implant (Eye disorders) | 3
White nodule on the prosthetic skirt (Eye disorders) | 1
left eye ocular pain (Eye disorders) | 1
fungal infection in the skirt of cornet artificial cornea (Eye disorders) | 1
abnormal serum enzyme levels (Eye disorders) | 1
elevated IOP (Eye disorders) | 1
eye pain (Eye disorders) | 1
watery eye (Eye disorders) | 1
Severe headache (crown top right) (General disorders) | 2 (3)
Light sensitivity (Eye disorders) | 1
nausea, body rash (General disorders) | 1
Pain around eye (Eye disorders) | 1
Choroidal Hemorrhage (Eye disorders) | 2
Vitreous Hemorrhage (Eye disorders) | 2
Shallow retinal detachment (Eye disorders) | 1
Hyphema (Eye disorders) | 1
Patient had vitrectomy, with PRP laser and Avastin injections done on July 28th due to the non-resol (Eye disorders) | 1
Dehiscence of prosthesis superiorly due to retraction (Eye disorders) | 1
Conjunctival retraction with dehiscence of prosthesis & possible corneal epithelial ingrowth (Eye disorders) | 1
During sep. of iris from cornea bleeding began & didnt allow surgeon to place device in good conditi (Eye disorders) | 1
Conjunctival retraction (Eye disorders) | 1
Disjunction of the nasal part of the KPRO (Eye disorders) | 1
Choroidal detachment and exudative detachment (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT04485858/Prot_000.pdf